CLINICAL TRIAL: NCT06687330
Title: Evaluating the Role of Step Counts in Predicting Readmission and Mortality in Unplanned Hospitalized Cancer Patients: A Prospective Observational Study, STEP-CANCER
Brief Title: Evaluating the Role of Step Counts in Predicting Readmission and Mortality
Acronym: STEP-CANCER
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, Medical Oncology Fellow, Gazi University
Other Study IDs: E-77082166-604.01-1070182
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-11

CONDITIONS: Exercise; Smart Watch; Quality of Life (QOL); Sleep Quality; Rehospitalization
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Tracking Mobility and Health Data with a Smartwatch in Discharged Oncology Patients to Predict Rehospitalization: A Prospective Study — The intervention involves daily monitoring of discharged oncology patients using a smartwatch (Huawei Watch Fit 2) to track physical activity (step count), heart rate, and sleep duration. Data is collected remotely via a smartphone app, allowing real-time tracking of health metrics post-discharge. This intervention is distinct in its focus on correlating mobility and physiological data with the risk of rehospitalization within a 30-90 day period. Patients will also receive recommendations to maintain daily walking routines as part of their post-discharge care. Additionally, quality of life and sleep quality assessments are conducted before discharge and at follow-up visits to provide a comprehensive overview of each patient's post-hospital recovery.

SUMMARY:
This study investigates the relationship between physical activity, heart rate, and sleep quality with recurrent hospitalizations among discharged oncology patients. Following discharge, patients will wear Huawei smartwatches to enable daily tracking of step count, heart rate, and sleep duration through a connected smartphone app. Patients will also complete the FACT Quality of Life Survey and the Pittsburgh Sleep Quality Index during follow-up visits. The smartwatch monitoring will occur during the first 30 days post-discharge, while overall patient follow-up will extend up to 90 days. This study aims to determine if lower levels of home mobility, as indicated by step count and other activity metrics, correlate with an increased risk of hospital readmission within the 30-90 day period.

DETAILED DESCRIPTION:
This observational study aims to investigate the relationship between post-discharge mobility metrics and the likelihood of recurrent hospitalizations among oncology patients. Eligible participants include those who have completed treatment in the oncology ward and have an ECOG performance status of 0-2. Patients admitted only for day treatments or with significant mobility limitations are excluded. Each patient receives a Huawei Watch Fit 2 smartwatch at discharge to record daily step counts, heart rate, and sleep duration, monitored remotely through a smartphone application.

In addition to these mobility and physiological metrics, patient-specific factors-such as diagnosis, reason for admission, date of last treatment, cancer stage, and age-are collected, as these may influence follow-up outcomes. Participants complete the FACT Quality of Life Survey and the Pittsburgh Sleep Quality Index at two time points: prior to discharge and again at follow-up, enabling a comparative assessment of quality of life and sleep quality over time. All patients receive general walking recommendations to support their recovery.

During the first 30 days post-discharge, activity and physiological data are continuously monitored through the app. The follow-up period extends to 90 days, during which any hospital readmissions are recorded. By analyzing trends in step count, sleep patterns, and heart rate variability, the study aims to determine whether decreased home mobility is associated with a higher risk of readmission, potentially enabling earlier interventions for at-risk individuals.

Participant recruitment for this study was completed ahead of schedule due to a higher-than-anticipated rate of eligible patient enrollment. The study is currently in the follow-up phase, and data collection for outcome measures is ongoing. The anticipated primary completion date is June 15, 2025.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older.
* Oncology Ward Discharge: Patients who have been discharged from the oncology ward following inpatient treatment.
* Cancer Diagnosis: Patients diagnosed with any form of cancer who received treatment in the oncology ward.
* Treatment Completion: Patients who have completed their scheduled inpatient oncology treatment and have been discharged.
* Performance Status: Patients with an ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2, indicating they are ambulatory and capable of basic physical activity.
* Follow-Up Availability: Patients who are willing and able to participate in a 90-day follow-up period after discharge.
* Technology Compliance: Patients who agree to wear a Huawei Watch Fit 2 smartwatch for the first 30 days post-discharge to track daily step count, heart rate, and sleep duration, and have access to a compatible smartphone for remote data monitoring.
* Survey Participation: Patients willing to complete the FACT Quality of Life Survey and Pittsburgh Sleep Quality Index before discharge and during follow-up visits.

Exclusion Criteria:

* Day Treatment Admissions: Patients admitted exclusively for day treatments or outpatient procedures, lacking a full inpatient admission in the oncology ward.
* Severe Mobility Limitations: Individuals with substantial mobility impairments, rendering them unable to perform basic ambulatory activities such as walking.
* Incompatibility with Technology Requirements: Patients who are unable or unwilling to wear the Huawei Watch Fit 2 smartwatch for data collection purposes or who lack access to a compatible smartphone for remote monitoring.
* Non-Adherence to Follow-Up Protocol: Patients who are unwilling or unable to comply with the 90-day follow-up requirements post-discharge.
* Incomplete Oncology Treatment Course: Individuals who have not completed the intended course of oncology treatment within the oncology ward prior to discharge.
* Cognitive or Psychiatric Impairments: Patients with significant cognitive or psychiatric disorders that impair their ability to provide informed consent or adhere to study protocols.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes oncology patients discharged from the inpatient ward after completing their treatment regimen. Eligible participants are adults (≥18 years) with various cancer types and an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2, indicating the ability to perform basic ambulatory activities. The cohort will be analyzed for the relationship between post-discharge physical activity-assessed through daily step counts, heart rate, and sleep duration-and the risk of readmission within 90 days. Exclusion criteria include patients with significant mobility limitations, cognitive or psychiatric impairments, or those admitted only for outpatient or same-day treatments.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Association Between Daily Step Count and Recurrent Hospitalization | 6 months
  To evaluate the relationship between daily step count, as recorded by a smartwatch, and the incidence of recurrent hospitalizations within 30 to 90 days post-discharge among oncology patients. The study aims to determine if lower daily step counts are associated with an increased risk of rehospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Nuriye Ozdemir, Prof. Dr., Study Chair — Gazi University; Osman Sutcuoglu, Associate Professor, Study Director — Ankara Etlik City Hospital; Orhun Akdogan, MD, Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara, Yenimahalle
  - Gazi University, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and in alignment with ethical guidelines protecting participant confidentiality. Data sharing is restricted to maintain compliance with institutional and national regulations governing patient privacy. Currently, no plans exist to provide IPD access beyond the research team responsible for the study.